CLINICAL TRIAL: NCT05533437
Title: Effect of Different Duration of Dry Needling on Muscles Strength of Flexor Forearm Muscles of Dominant Hand in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Responsible Party: Principal Investigator, faizan kashoo, PT, Lecturer, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AIHMS-2 New Delhi
Record Dates: First submitted 2022-09-06; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Dry Needling
Keywords: dry needling; kinesio tapping; Healthy adults
MeSH Terms: interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): During dry needling, a practitioner inserts several filiform needles into your skin. Filiform needles are fine, short, stainless steel needles that don't inject fluid into the body.
  Interventions: Device: dry needling
- kinesio taping (Active Comparator): The Kinesio Taping Method is a therapeutic taping technique which alleviates pain and facilitates lymphatic drainage by microscopically lifting the skin. This lifting affect forms convolutions in the skin increasing interstitial space and allowing for decreased inflammation in affected areas. Based upon research and years of clinical use, The Kinesio Taping Method specifically applies Kinesio tape based on evaluation and assessment to dictate a specific application.
  Interventions: Other: kinesio taping

INTERVENTIONS:
Device: dry needling — the dry needle inserted to area of pain
  Arms: Dry needling
Other: kinesio taping — kinesio taping
  Arms: kinesio taping

SUMMARY:
Dry needling is typically used to treat muscles, ligaments, tendons, subcutaneous fascia, scar tissue, peripheral nerves, and neurovascular bundles for the management of a variety of neuromusculoskeletal pain syndromes.However, there are contradictory research articles about the optimal duration of dry needling per session.

DETAILED DESCRIPTION:
Dry needling is 'an invasive technique used by physical therapists to treat myofascial pain that uses a dry needle, without medication or injection, which is inserted into areas of the muscle known as trigger point defines dry needling as including both muscular and connective tissues, but not neural stimulation. The paper reads, 'dry needling is a skilled intervention that uses a thin filiform needle to penetrate the skin and stimulate underlying myofascial trigger points, muscular, and connective tissues for the management of neuromusculoskeletal pain and movement impairments.

The dry needling is reported to improve the level of pain, muscle strength, and flexibility. However, the optimal duration of dry needling to improve muscle strength is still Unknown.

ELIGIBILITY:
Inclusion Criteria:

Patient with osteoarthritis

Exclusion Criteria:

Patient with musculoskeletal disorders Metabolic disorders causing knee pain Surgery

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Level of pain on pain scale | 3 months
  Level of pain in the pain scale

CONTACTS AND LOCATIONS:
Locations (1):
- AIMHS, New Delhi, India